CLINICAL TRIAL: NCT05490914
Title: The Prognostic Factors of COVID-19 ARDS Patients and Their Long-term Follow-up of Pulmonary Function Test
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005059RIND
Record Dates: First submitted 2022-04-20; First posted 2022-08-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19; ARDS; Lung mechanics; Ventilation strategy; Lung mechanics&function
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: COVID-19 case
- Control Group: Healthy population without COVID-19

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is an emerging infectious disease with high transmissibility. Around 20-25% of infected individuals develop severe COVID-19 disease requiring hospitalization and 5-8% require intubation secondary to viral pneumonia and acute respiratory distress syndrome (ARDS). Distinct features of COVID-19 ARDS were found since Nov 2019, including relatively normal lung mechanics, activation of the RAAS system, selective injury of type II alveolar cells, and presence of vasodilation vessel and micro-thrombosis. The mechanism, potential useful biomarker, and the optimal ventilation strategies for COVID-19 ARDS need to be systematically studied. This study hypothesized that the low-tidal volume ventilation strategy is effective in COVID-19 ARDS. We will retrospectively review the clinical presentation, epidemiologic data, laboratory and image examination, medication use, lung mechanics、serum biomarker, long-term pulmonary function test, and clinical outcomes in COVID-19 ARDS, influenza ARDS, and SARS ARDS patients. We will also prospectively monitor the lung function of COVID ARDS patients using personal pulmonary function devices after discharge from NTUH. The overall purpose of this study is to investigate the prognostic indicators of COVID ARDS patients and their long-term pulmonary function follow-up.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is an emerging infectious disease with high transmissibility. Around 20-25% of infected individuals develop severe COVID-19 disease requiring hospitalization and 5-8% require intubation secondary to viral pneumonia and acute respiratory distress syndrome (ARDS). Distinct features of COVID-19 ARDS were found since Nov 2019, including relatively normal lung mechanics, activation of the RAAS system, selective injury of type II alveolar cells, and presence of vasodilation vessel and micro-thrombosis. The mechanism, potential useful biomarker, and the optimal ventilation strategies for COVID-19 ARDS need to be systematically studied. This study hypothesized that the low-tidal volume ventilation strategy is effective in COVID-19 ARDS. We will retrospectively review the clinical presentation, epidemiologic data, laboratory and image examination, medication use, lung mechanics、serum biomarker, long-term pulmonary function test, and clinical outcomes in COVID-19 ARDS, influenza ARDS, and SARS ARDS patients. We will also prospectively monitor the lung function of COVID ARDS patients using personal pulmonary function devices after discharge from NTUH. The overall purpose of this study is to investigate the prognostic indicators of COVID ARDS patients and their long-term pulmonary function follow-up.The SARS-CoV-2 (COVID-19) ARDS is an emerging novel devastating disease with high mortality. Distinct features were found since Nov 2019, including relatively normal lung mechanics, activation of the RAAS system, selective injury of type II alveolar cells, and presence of vasodilation vessel and micro-thrombosis. The optimal ventilation strategies for COVID-19 ARDS need to be systematically studied. The overall purpose of this study is to investigate the prognostic indicators in COVID-19 ARDS patients.Specific Aim 1: To develop a REDcap database of clinical and biologic information in subjects with COVID-19, and to investigate the prognostic indicators compared with influenza and SARS ARDS patients.Specific Aim 2: To follow up the long-term change pulmonary function test of COVID ARDS patients using home-based personal pulmonary function test device

ELIGIBILITY:
Inclusion Criteria:

1. Adult >20 years old
2. Retrospective cohort by medical chart review：COVID-19 patients, Influenza patients, and SARS patients at NTUH
3. Prospective cohort：COVID-19 confirmed patients intubated and receiving mechanical ventilation > 24 hours at NTUH, got extubated and discharged

Exclusion Criteria:

1. Pregnancy
2. No consent/inability to obtain consent or appropriate legal representative not available

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experimental Group：COVID-19 case
  Control Group：Healthy population without COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome of the retrospective cohort | on ventilation day 28
  liberation from mechanical ventilation/ventilator dependency on ventilation day 28
Primary Outcome of the retrospective cohort | through study completion, an average of 1 year
  ICU and in-hospital mortality

SECONDARY OUTCOMES:
Outcome of the prospective cohort: pulmonary function test will be performed daily by the patients after discharge from NTUH | through study completion, an average of 1 year
  forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC)

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan